CLINICAL TRIAL: NCT04930302
Title: Optimizing the Pharmacotherapy of Vascular Surgery Patients at Hospital Admission, at Discharge and at Post-discharge Check-up: Quasi-experimental Clinical Uncontrolled Trial (PHAROS)
Acronym: PHAROS
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Slovakia (Other)
Responsible Party: Principal Investigator, Slavka Porubcova, PharmDr., Principal Investigator, National Institute of Cardiovascular Diseases, Slovakia
Other Study IDs: PHAR008NUSCH
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Medication Errors and Other Product Use Errors and Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to assess the impact of pharmaceutical care in collaboration with physicians on prevalence of DRPs at hospital admission and discharge in patients with carotid artery disease or lower extermity artery disease hospitalized at the Department of Vascular Surgery.

The key focus area of this project will be the identification of DRPs, their occurrence and type. As a part of further research, the investigators want to analyze the a) acceptance rate of pharmaceutical intervention by physicians. Proportion of accepted interventions by physicians was calculated and b) patients' understanding of his/her pharmacotherapy assessed on a three-point scale at hospital admission.

Hypothesis:

Null hypothesis: Pharmaceutical care provided at hospital admission and at hospital discharge does not reduce prevalence rates of DRPs in patients with carotid artery disease or lower extermity artery disease hospitalized at the Department of Vascular Surgery.

Alternative hypothesis: Pharmaceutical care provided at hospital admission and at hospital discharge reduces prevalence rates of DRPs in patients with carotid artery disease or lower extermity artery disease hospitalized at the Department of Vascular Surgery.

Primary outcomes:

Change in the prevalence rate of DRPs at hospital admission vs. hospital discharge.

Secondary outcomes:

1. acceptance rate of pharmaceutical intervention by physician
2. patients' understanding of his/her pharmacotherapy

DETAILED DESCRIPTION:
Medication reconciliation, medication review and patient education performed by a trained pharmacist in two timepoints.

All comments with a proposal from the pharmacist will be recorded in written together with a record of the therapy, entered in the patient's medical record and communicated with the physician.

Timepoints for intervention:

1. At hospital admission

   The patient is normally admitted to the planned hospitalization by the physician in cooperation with the nurse as described above. If the patient is over 18 years of age, takes more than three medicines, speaks and understands Slovak language and has signed an informed consent to participate in biomedical research, after being placed in a bed, a pharmacist comes to the patient and performs MR. During MR, the pharmacist creates a record of the patient's therapy (MR form for admission - attachment No. 2), the original of which is placed in the patient's medical record, and a copy is placed to pharmacist´s records.

   Steps in MR:
   1. As part of the invitation to hospitalization (by telephone, in writing), the patient will be asked to bring all their medications and a complete medication list, which will be used in consultation with the pharmacist regarding their proper use.
   2. Completion of BPMH

      BPMH is a treatment overview obtained by a healthcare professional that contains all the medicines (prescription medicines and over-the-counter drugs) that the patient is taking, using various sources of information. The source of information can be a drug record, an admission report and a course, historical records from the HIS, information from the patient or his family member. BPMH is different and more complex than the routine history of primary treatment (which is often a rapid history of patient treatment). The BPMH includes the name of the medicine, the dose, the frequency and the route of the medicines that the patient is currently taking, although it may differ from what was actually written in the drug list.

      The types of drugs that need to be recorded for BPMH include:
      * prescription drugs
      * over-the-counter drugs
      * nutritional supplements
      * herbal medicines, medicinal teas
      * recreational drugs
      * regular consumption of certain foods (e.g. grapefruit)
      * special emphasis should be placed on specific forms of medicines such as inhalers, eye drops, topical semi-solid medicines, or medicines taken every few weeks (bisphosphonates)

      One of the recorded parameters is patient understanding. It is evaluated in three steps - the patient knows / does not know the name of the drug (1/0), the patient knows / does not know the indication of the drug (1/0) and the patient knows / does not know the dosage of the drug (1/0).

      If the patient is unable to attend the interview, other sources may be used to obtain a medical history or to clarify conflicting information. Other resources should never be a substitute for a thorough conversation with the patient and / or family members.
   3. Verification and documentation of BPMH

   Medicinal product information should be verified by more than one other source. Sources for the initial acquisition of an overview of pharmacotherapy are the admission report, the history of hospitalization, outpatient reports, HIS, the course at admission. The investigators verify the information obtained by speaking with a patient or his family member, the provided drug list or drugs.

   Within the WHO SOP, the investigators chose a retroactive MR model at admission for our biomedical research. In a retroactive model, in accordance with the method described above, the patient is admitted by a physician in cooperation with a nurse by default, and a drug course is created, a daily prescription of drugs for the patient. In this case, the BPMH is determined after admission by a physician / nurse.

   The result of Part b) is a comparison of prescribed and actually used medicines to patients (BMPH) with marked discrepancies.

   Medication review with pharmaceutical intervention at patient admission The basis for performing patient therapy optimization is the acquisition of BPMH and patient factors such as the reason for hospitalization, current health status, comorbidities, height, weight, heart rate, blood pressure and the results of examinations of biochemical and hematological parameters.

   The detected BPMH is written to the case report form (CRF) (attachment No. 4) . It is then analyzed in the context of the patient's overall health condition and DRPs are identified. Each detected discrepancy is assigned an alphanumeric code according to the PCNE V9.00 classification. The patient's personal data is anonymized.

   Discrepancies in therapy should be consulted with the treating physician within 24 hours of admission.

   Evaluation of therapy based on DRPs and PCNE classification After receiving BPMH and a detailed study of the reason for hospitalization, current medical condition, and any comorbidities of the patient, the pharmacist draws information about the patient's weight, height, heart rate, and blood pressure from the admission report. Subsequently, he/she studies the results of biochemical and hematological examinations. The pharmacist focuses on the results of examinations related to pharmacotherapy and the determination of the function of elimination organs. These are mainly the serum potassium, serum creatinine, serum uric acid, liver transaminases, lipidogram, C-reactive protein. Renal function is calculated based on the Cockcroft and Gault creatinine clearance estimate and the CKD-EPI glomerular filtration rate estimate. From the hematological results, the pharmacist focuses on INR, aPTT-R, anti Xa activity, platelet count and others.

   The pharmacist controls duplication in the drugs used; the indications of the drugs used according to the patient's comorbidities; compliance with the maximum recommended doses of drugs according to the SPC; the suitability of the choice of dosage form; drug interactions using the computerized interaction database, the LexiComp℗, SPC, pharmacological findings, published scientific papers and case reports; newly manifested adverse drug reactions.
2. At hospital discharge

The pharmacist performs a MR when discharging a patient from the hospital, similar to the admission. MR form for discharge is used (attachment No. 5). When evaluating a patient's pharmacotherapy on discharge from hospital, the BPMH obtained at the patient's admission will be used as a source of information. The BPMH is then compared with the list of medicines that are recorded in the release report. The pharmacist will compare the two lists of medicines, focusing on the identification of DRPs with special regard to the re-introduction of the chronic therapy which the patient was taking before coming to the hospital. As part of this research, the pharmacist will meet with the patient during his discharge from the hospital and discuss with him the management of his further pharmacotherapy. Pharmacists provide an understandable summary list of patient's medicines explaining importance and the correct use of medicine (attachment No. 6).

Medication review with pharmaceutical intervention at patient discharge The pharmacist analyzes pharmacotherapy in the context of the patient's state of health and the results of laboratory tests, similar to the patient's admission as described above. Detected DRPs are then consulted with the treating physician and recorded in the CRF.

The result of the pharmacist's intervention at discharge is the completion of the MR form for discharge and the writing of all comments on pharmacotherapy in the form of a summary report. Discrepancies and comments are consulted with the physician.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the date of admission for hospitalization
2. patients taking at least 3 medications
3. patients with carotid artery disease or lower extremity artery disease

Exclusion Criteria:

1. Acute patients.Due to the urgent health condition, medication reconciliation is not the priority in these patients, furthermore, rendering the BPMH collection impossible.
2. Patients transferred from other hospitals/wards
3. Not willing to sign the informed consent form for the study
4. Not understanding Slovak language
5. Presence of any mental disorder affecting memory and recall ability (such as Alzheimer's disease)
6. Any other reason at the discretion of the investigator why he/she deems the participant not eligible for study participation (all such reasons will be recorded)
7. Participation in another clinical study
8. Furthermore, patients transferred to other hospitals/wards will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years of age) Vascular surgery patients with carotid artery disease or lower extremity artery disease admitted for hospitalization at the study setting during the course of the study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in prevalence rate of drug related problems | through study completion, an average of 1 year
  Change in the prevalence rate of drug related problems at a) hospital admission vs. hospital discharge, b) hospital discharge vs. post-discharge check-up.

SECONDARY OUTCOMES:
patients characteristics | through study completion, an average of 1 year
  weight in kilograms
patients characteristics | through study completion, an average of 1 year
  height in meters
patients characteristics | through study completion, an average of 1 year
  diagnosis
patients characteristics | through study completion, an average of 1 year
  biochemical and hematological parameters (levels of Na+, K+, Cr, CKD-EPI, platelet levels)
patients characteristics | through study completion, an average of 1 year
  age
patients characteristics | through study completion, an average of 1 year
  sex
patients characteristics | through study completion, an average of 1 year
  social and employement status
patients characteristics | through study completion, an average of 1 year
  level of understanding of used pharmacotherapy
Medication characteristics | through study completion, an average of 1 year
  name of drug/medicine
Medication characteristics | through study completion, an average of 1 year
  ATC of drug
Medication characteristics | through study completion, an average of 1 year
  dose
Medication characteristics | through study completion, an average of 1 year
  dosage form of medicine
Medication characteristics | through study completion, an average of 1 year
  frequency of using

CONTACTS AND LOCATIONS:
Overall Officials: Slavka Porubcova, PharmDr., Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases, Slovakia, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porubcova S, Lajtmanova K, Szmicsekova K, Slezakova V, Tomka J, Tesar T. Optimizing the Pharmacotherapy of Vascular Surgery Patients at Hospital Admission and Discharge (PHAROS): Protocol for a Quasi-Experimental Clinical Uncontrolled Trial. JMIR Res Protoc. 2025 Mar 19;14:e60728. doi: 10.2196/60728. PMID 40106812
- [Derived] Porubcova S, Szmicsekova K, Lajtmanova K, Slezakova V, Jakubik M, Drobna E, Tomka J, Kobliskova Z, Masarykova L, Lehocka L, Tesar T. Pharmacist-led interventions for vascular surgery patients: a prospective study on reducing drug-related problems. BMC Health Serv Res. 2024 Dec 18;24(1):1564. doi: 10.1186/s12913-024-12015-7. PMID 39695586